CLINICAL TRIAL: NCT03409211
Title: Patterns After Administration of MCFAs in Psoriasis and Psoriatic Arthritis
Acronym: PAMPPA
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-00748
Record Dates: First submitted 2018-01-05; First posted 2018-01-24 (Actual); Last update posted 2020-12-02 (Actual); Status verified 2020-12

CONDITIONS: Psoriasis; Psoriatic Arthritis
MeSH Terms: conditions — Psoriasis; Arthritis, Psoriatic | interventions — Coconut Oil; Dietary Supplements

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Pso (Active Comparator): with or without PsA
  Interventions: Dietary Supplement: PEVCO; Dietary Supplement: Dietary Supplement Capsules without Coconut Oil
- Healthy Subjects (Active Comparator): Without PsA
  Interventions: Dietary Supplement: PEVCO; Dietary Supplement: Dietary Supplement Capsules without Coconut Oil

INTERVENTIONS:
Dietary Supplement: PEVCO — All subjects will receive PEVCO for 6 more weeks.
  Other Names: Coconut Oil
Dietary Supplement: Dietary Supplement Capsules without Coconut Oil — All subjects will receive placebo (PBO) for 3 weeks

SUMMARY:
This is a proof-of-principle, placebo-controlled, open label study to assess the improvement in the Treg counts and PASI Scores with PEVCO given at 1000 mg four times daily in patients with PsO (subjects may or may not have PsA) , who have active disease and are not currently receiving other therapy (as defined by the inclusion/exclusion criteria) compared to healthy subjects.

The patients and healthy controls will receive placebo or PEVCO for a total of 9 weeks (3 weeks for placebo, followed by 6 weeks for PEVCO). No topical or systemic medications will be used during this period.

ELIGIBILITY:
Inclusion Criteria:

* Have an active [psoriatric plaque >2cm

Exclusion Criteria:

* History of sensitivity to study compound or any of their excipients
* Previous intolerance to PEVCO or related compounds
* Current (within 3 months of screening) treatment with DMARDs
* Current (within 3 months of screening) treatment with biologic therapies (including but limited to anti-TNF,anti-IL-17, anti-IL-12/23)
* Current antibiotic treatment (within 3 months of screening)
* current consumption of probiotics (within 3 months of screening)
* Severe hepatic impairment (eg, ac-sites and/or clinical signs of coagulopathy)
* Renal failure (eGFR ,30 or require dialysis) by history
* History of other autoimmune or inflammatory skin disease
* Current immunodeficiency state (cancer, HIV, others)
* Current immunodeficiency state (cancer, HIV, Other)
* Concern for inability of the patient to comply with study procedure, and or follow up (alcohol or drug abuse)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2017-12-12 (Actual); Primary Completion 2019-09-30 (Actual); Study Completion 2019-09-30 (Actual)

PRIMARY OUTCOMES:
Change in % of Treg Cells in Blood | 6 Weeks
  % change in the expansion of regulatory T cells; demonstrate an increase in %Treg at 6 weeks.

SECONDARY OUTCOMES:
Increase in Medium Chain Fatty Acids (MCFA) content in the stool | 12 Weeks
  Change in the amount of MCFA in stool
Improvement in skin disease severity PASI scores 50 | 12 Weeks
  indicating 50% reduction in psoriasis
Improvement in skin disease severity PASI scores 75 | 12 Weeks
  indicating 75% reduction in psoriasis
Improvement in skin disease severity PASI scores 90 | 12 Weeks
  indicating 90% reduction in psoriasis
Improvement in the tender joint/swollen joint (TJ/SJ) counts at 6 weeks. | 6 Weeks
  To assess whether PEVCO 1000 mg four times daily for 6 weeks improves:
  * 66/68 Tender-joint count
  * 66/68 Swollen-joint count

CONTACTS AND LOCATIONS:
Overall Officials: Jose Scher, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided